CLINICAL TRIAL: NCT02951559
Title: Study of Nasal Brushing Collected OLFActory MUcosa Samples in the Diagnosis of Human Encephalopathies
Brief Title: SOLFAMU Study of Nasal Brushing Collected OLFActory MUcosa Samples in the Diagnosis of Human Encephalopathies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Di Perri, Professor of Infectious Diseases, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOLFAMU
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Encephalopathy; HIV-encephalopathy; Alzheimer Dementia
MeSH Terms: conditions — Brain Diseases; AIDS Dementia Complex; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Diagnostic study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brushing (Experimental): Patients will undergo nasal brushing as further described additionally to other gold standard practices according to the suspected aetiology (brain MRI, lumbar puncture, plasma tests, etc.)
  Interventions: Device: Nasal Brushing

INTERVENTIONS:
Device: Nasal Brushing — Nasal brushing will be performed in non-sedated patients as follows. After administration of a local vasoconstrictor (1% epinephrine) with the use of a nasal tampon, inserted into the nasal cavity of the patient to locate the olfactory mucosa lining the nasal vault. A sterile, disposable brush ("Copanflock", "Copan", Brescia, Italy) will be inserted gently rolled on the mucosal surface, withdrawn,and immersed in 0.9% saline solution, UTM (Universal Transporter Medium) or 4% formaldehyde. Two swabs will be collected for each nostril.

SUMMARY:
Encephalopathies are a group of central nervous system (CNS) affection with heterogeneous etiology. Several causes have been recognized including neurodegenerative, vascular, infectious, autoimmune, toxic or allergic affections or secondary to systemic disorders. While 30-50% of acute encephalitis remains without etiological definition, definitive criteria for neurodegenerative diseases are usually unavailable in vivo and possible or probable definitions are used. The Olfactory mucosa (OM) is the part of the nasal mucosa that carries the specialized sensory organ for the modality of smell; the olfactory epithelium is composed of five principal cell types including olfactory receptor neurons. A sample of OM may be collected through a rhinoscopy-guided brushing: it is well-accepted by patients, not-contraindicated in patients with raised intracranial pressure and associated with almost no side-effects. Nasal brushing has recently been proposed for the in vivo diagnosis of Creutzfeldt-Jakob disease (CJD).

Aims of the project are:

1. Training of ear throat and nose (ETN), Infectious disease (ID) and neurology (NEU) specialists in the technique of nasal brushing;
2. Conducting a prospective study comparing the use of nasal brushing with gold-standard criteria in the diagnosis of Encephalopathies;
3. Increasing the diagnostic and prognostic power in the diagnosis of encephalopathies.

A prospective, case control, multicentric study enrolling 400 patients and 100 controls (patients with nasal stenosis undergoing rhinoscopy for clinical reasons). Patients will be diagnosed and followed according to international guidelines and local clinical practice. Cerebrospinal fluid and magnetic resonance imaging will be used, where indicated, for the diagnosis according to the clinical or radiological suspect.

ELIGIBILITY:
Inclusion criteria for cases:

* age>18 years;
* signing a written informed consent (by the patients or his/her legal representant);
* clinical suspect of encephalopathy (acute or subacute) including acute encephalitis, neurodegenerative disorders and HIV-associated neurocognitive disorders.

Inclusion criteria for controls:

* age>18 years;
* signing a written informed consent (by the patients or his/her legal representant); • clinical indication for rhinoscopy for stenotic disease of nasal sept or turbinates.

Exclusion criteria:

* Nasal anatomical abnormalities precluding the execution of nasal brushing;
* Serious general conditions and/or comorbidities in patients for whom nasal brushing may be a risk factor precipitating their pre-existing condition;
* Anti-coagulant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-03; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic concordance with gold standard diagnostic procedures | Single-visit
  Positive and negative predictive values and correct classification rates of OM tests versus gold standard diagnostic procedures

SECONDARY OUTCOMES:
Side effects of the nasal brushing | Up to 6 months after the procedure
  Prevalence of side effects reported during the brushing and up to 6 months afterwards
Cytological and immunohistochemistry examination of nasal brushing smear (neuronal abnormalities and expression of specific markers according to the different aetiologies) | single-visit
  Prevalence of samples showing: abnormalities in cytological examination, antiOMP (Olfactory Marker Protein) positive cells, white blood cells and subtypes.
OM markers of neuronal damage and amyloid deposition | single-visit
  Quantification of tau, p-tau, 1-42 beta amyloid, S100beta, alpha synuclein, TDP-43 (TAR DNA-binding protein 43) on cell blocks and supernatant

CONTACTS AND LOCATIONS:
Overall Officials: GIOVANNI DI PERRI, MD, PhD, Principal Investigator — University of Torino
Locations (1):
- University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No